CLINICAL TRIAL: NCT03533712
Title: Effect of a Fortified Balanced Energy-Protein Supplement on Birth Outcome and Child Growth in Houndé District, Burkina Faso.
Acronym: MISAME-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); AfricSanté, Burkina Faso (Unknown); International Food Policy Research Institute (Other); University of California, Davis (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, VakgroepLevensmiddelentechnologieVoedselveiligheidGezondheid, Prof. dr. Patrick Kolsteren, University Ghent
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: OPP1175213
Record Dates: First submitted 2018-04-23; First posted 2018-05-23 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Small for Gestational Age at Delivery; Low Birth Weight; Prematurity; Infant Malnutrition
MeSH Terms: conditions — Premature Birth; Infant Nutrition Disorders | interventions — BEP protocol

STUDY DESIGN:
Intervention Model Description: The intervention study is a randomized controlled 2x2 factorial efficacy trial. At study inclusion, eligible pregnant women will be randomly assigned to the prenatal intervention or control group, and randomly assigned to a postnatal intervention or control group. The intervention group will receive daily a fortified BEP supplement to be consumed under supervision for the duration of pregnancy/lactation. Both control and intervention group will receive the standard iron and folic acid tablet through the regular ante natal care program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fortified BEP supplement (Experimental): Intervention: Dietary Supplement: Fortified balanced energy-protein (BEP) supplement + iron and folic acid supplement.
  Interventions: Dietary Supplement: Fortified balanced energy-protein (BEP) supplement
- Fe and folic acid (Active Comparator): Dietary Supplement: Fe and folic acid supplement.
  Interventions: Dietary Supplement: Fe and folic acid supplement

INTERVENTIONS:
Dietary Supplement: Fortified balanced energy-protein (BEP) supplement — The product contains the following target nutrients:
  * Total energy: 250-500 kcal per daily serving
  * Fat content: 10-60% of energy intake
  * Protein content: 16 g (range 14-18 g) with a Digestible Indispensable Amino Acid Score (DIAAS) of ≥ 0.9
  * Carbohydrate (CHO) Content: no specific recommendations, relative to fat and protein content.
  * Trans Fats: <1% energy intake Micronutrients include the following: A, D, E, K, B1 (thiamin), B2 (riboflavin), B3 (niacin), B6 (pyridoxine), B9 (folate), B12 and C; minerals: iron, zinc, iodine, calcium, phosphorous, copper, and selenium.
  The final composition of macro en micronutrients will be available after the acceptability testing (phase 1) and will be determined by 1) the product type and 2) the preferred taste.
  Arms: Fortified BEP supplement
Dietary Supplement: Fe and folic acid supplement — Routine iron and folic acid supplementation.
  Arms: Fe and folic acid

SUMMARY:
The 2016 WHO antenatal care guidelines stated that pregnant women in undernourished populations should receive fortified balanced energy-protein (BEP) supplements to reduce the risk of stillbirth and small-for-gestational-age birth. However, acceptable supplements and delivery channels must be determined for different contexts.

The present proposal therefore will 1) perform a formative study to identify the most suitable (acceptability and utilization) BEP supplement for pregnant women in rural Burkina Faso (phase 1) and 2) evaluate the efficacy of this supplement to improve birth weight, fetal and infant growth (phase 2). The nutritional composition of the BEP supplement was established during an expert convening at the BMGF in September 2016. Private sector partners will prepare the supplements in the selected forms with the recommended nutrient composition.

DETAILED DESCRIPTION:
Pregnancy remains a challenging period in the life of many women in low- and middle-income countries. Maternal mortality remains high and many newborns suffer from premature delivery and /or gestational growth retardation both in length and in weight accumulation.

The 2016 WHO antenatal care guidelines stated that pregnant women in undernourished populations should receive fortified balanced energy-protein (BEP) supplements to reduce the risk of stillbirth and small-for-gestational-age birth. However, acceptable supplements and delivery channels must be determined for different contexts.

The purpose of this study is to assess the efficacy of a fortified BEP supplement for pregnant and lactating women to improve birth weight, fetal and infant growth.

This research includes 2 phases:

* Phase 1 - part 1: Formative research to identify preferred product types of a fortified BEP supplement;
* Phase 1 - part 2: Formative research with a 10-week home-feeding trial to determine the acceptability of a fortified BEP supplement for longer-term consumption.
* Phase 2: A community-based, individually randomized efficacy trial of the fortified BEP food supplement including 1,776 pregnant and lactating women aimed at testing 2 hypothesis: supplementing pregnant and lactating women with a fortified BEP supplement will improve fetal growth; improving fetal growth will have a positive effect on health and growth during infancy.

ELIGIBILITY:
Inclusion Criteria:

* Participant age (15-40 years).
* Pregnant as determined by a pregnancy test and confirmed by ultrasound.
* Women who signed the informed consent form (in case of minors the parents or husband signs)

Exclusion Criteria:

* Women planning to leave the area before delivery.
* Women who plan to deliver outside the area.
* Pregnancies with a gestational age > 20 weeks at study inclusion.
* Women with multi-fetal gestation (exclusion from analysis).
* Women who are allergic to peanuts.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1788 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Small-for-Gestational-age (SGA) | within 72h after birth
  Incidence of Small-for-Gestational-age (SGA) defined as <10th centile of birthweight for gestational age standard, InterGrowth 21st reference.
Length-for-age Z-scores (LAZ) | at 6 months (and 12 months on a subsample)
  Mean of Length-for-Age Z-scores (LAZ), WHO multi-country reference.

SECONDARY OUTCOMES:
Birth weight | within 72h after birth
Birth length | within 72h after birth
Chest circumference | within 72h after birth
Head circumference | within 72h after birth
Mid-upper arm circumference | within 72h after birth
Gestational age | at delivery
Preterm birth | at delivery
  Incidence of preterm birth at <37 weeks of gestation
Large-for-gestational age | within 72h after birth
  Defined as a birth weight ≥90th centile intergrowth 21st reference
Ponderal or Rohrer's index' | within 72 hours after birth
  Defined as birth weight/birth length3
Fetal loss | during pregnancy
  Fetal death at <24 completed weeks of gestational age
Stillbirths | during pregnancy
  Fetal death at ≥ 24 weeks gestational age
Neonatal mortality | between birth and ≤ 28 days of life
  (1) Early neonatal mortality: deaths between birth and ≤ 7 days of life; (2) Neonatal mortality: deaths between birth and ≤28 days of life; (3) Late neonatal mortality deaths between >7 days and ≤28 days of life
Prenatal weight gain | between study inclusion until just before delivery
  Weight change between study inclusion until just before delivery: total and trimester specific
Gestational weight change | between study inclusion until 1 month after delivery
  Difference in maternal weight between maternal weight one month after delivery and maternal weight at study inclusion
Probable and possible maternal postnatal depression | (1) at 2 months of child age; (2) at 6 months of child age
  Measured using the 10-item Edinburgh postnatal depression scale. Probable depression is defined as EPDS>12. Possible depression is defined as EPDS>9 .
Women's minimum and mean dietary diversity score | from study inclusion until delivery
  Measured biweekly using the 10 food group indicator as proposed by FAO. Minimum dietary diversity is defined as having consumed at least 5 food groups over the last 24 hours.
Maternal anemia | at the third antenatal consultation
  Hemoglobin concentration <11g/dL
Weight-for-Age Z-score | at 6 months of age
  WAZ, calculated using the WHO growth reference
Weight-for-Length Z-score | at 6 months of age
  WLZ, calculated using the WHO growth reference
Stunting | at 6 months of age
  Length-for-Age Z-score (LAZ) <-2, calculated using the WHO growth reference
Wasting | at 6 months of age
  Weight-for-Length Z-score (WLZ) <-2, calculated using the WHO growth reference
Underweight | at 6 months of age
  Weight-for-Age Z-score (WAZ) <-2, calculated using the WHO growth reference
Incidence of child wasting | over first 6 months of life
Child weight gain | over first 6 months of life
  Monthly change in child weight
Monthly change in LAZ | over first 6 months of life
Monthly change in WHZ | over first 6 months of life
Monthly change in WAZ | over first 6 months of life
Monthly change in head circumference | over first 6 months of life
Exclusive breastfeeding | during the first 6 months of life
  Duration of exclusive breastfeeding
Child mortality | between birth and 6 months of age
Child morbidity symptoms | over first 6 months of life
  Signs include fever, vomiting, diarrhea, cough, difficult breathing, running nose
Child anemia | at 6 months of age
  Hemoglobin concentration <11g/dL
Hemoglobin concentration | at 6 months of age
Infant body composition | first 3 months of life
  Sub-sample
Maternal body composition | first 3 months after delivery
  Sub-sample
Breast milk composition | between 1-2 and 3-4 months
  Sub-sample
Relative average telomere length | At birth
  The umbilical cord blood will be analyzed to verify telomere length using qPCR on a sub-sample. Telomere lengths will be expressed as the ratio of telomere copy number to single-copy gene number (T/S) relative to the mean T/S ratio of the entire sample.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kolsteren, Prof. dr., Study Chair — University Ghent; Carl Lachat, Prof. dr., Study Director — University Ghent; Katrien W Vanslambrouck, MD, Principal Investigator — University Ghent; Brenda PH de Kok, MSc., Principal Investigator — University Ghent; Lieven F Huybregts, PhD, Principal Investigator — IFPRI; Laeticia Celine Toe, MD MSc., Principal Investigator — IRSS; Sheila Isanaka, Asst. Prof., Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Houndé district, Houndé, Tuy, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Share study data with a similar study ongoing in Nepal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Argaw A, Toe LC, Hanley-Cook G, Dailey-Chwalibog T, de Kok B, Ouedraogo L, Compaore A, Ouedraogo M, Sawadogo A, Ganaba R, Vanslambrouck K, Kolsteren P, Lachat C, Huybregts L. Effect of prenatal micronutrient-fortified balanced energy-protein supplementation on maternal and newborn body composition: A sub-study from the MISAME-III randomized controlled efficacy trial in rural Burkina Faso. PLoS Med. 2023 Jul 24;20(7):e1004242. doi: 10.1371/journal.pmed.1004242. eCollection 2023 Jul. PMID 37486952
- [Derived] Argaw A, de Kok B, Toe LC, Hanley-Cook G, Dailey-Chwalibog T, Ouedraogo M, Compaore A, Vanslambrouck K, Ganaba R, Kolsteren P, Lachat C, Huybregts L. Fortified balanced energy-protein supplementation during pregnancy and lactation and infant growth in rural Burkina Faso: A 2 x 2 factorial individually randomized controlled trial. PLoS Med. 2023 Feb 6;20(2):e1004186. doi: 10.1371/journal.pmed.1004186. eCollection 2023 Feb. PMID 36745684
- [Derived] Hanley-Cook G, Toe LC, Tesfamariam K, de Kok B, Argaw A, Compaore A, Ouedraogo M, Dailey-Chwalibog T, Kolsteren P, Lachat C, Huybregts L. Fortified Balanced Energy-Protein Supplementation, Maternal Anemia, and Gestational Weight Gain: A Randomized Controlled Efficacy Trial among Pregnant Women in Rural Burkina Faso. J Nutr. 2022 Oct 6;152(10):2277-2286. doi: 10.1093/jn/nxac171. PMID 35906874
- [Derived] de Kok B, Toe LC, Hanley-Cook G, Argaw A, Ouedraogo M, Compaore A, Vanslambrouck K, Dailey-Chwalibog T, Ganaba R, Kolsteren P, Huybregts L, Lachat C. Prenatal fortified balanced energy-protein supplementation and birth outcomes in rural Burkina Faso: A randomized controlled efficacy trial. PLoS Med. 2022 May 13;19(5):e1004002. doi: 10.1371/journal.pmed.1004002. eCollection 2022 May. PMID 35560315
- [Derived] Hanley-Cook GT, Argaw A, de Kok B, Toe LC, Dailey-Chwalibog T, Ouedraogo M, Kolsteren P, Huybregts L, Lachat C. Seasonality and Day-to-Day Variability of Dietary Diversity: Longitudinal Study of Pregnant Women Enrolled in a Randomized Controlled Efficacy Trial in Rural Burkina Faso. J Nutr. 2022 Sep 6;152(9):2145-2154. doi: 10.1093/jn/nxac104. PMID 35524695
- [Derived] de Kok B, Argaw A, Hanley-Cook G, Toe LC, Ouedraogo M, Dailey-Chwalibog T, Diop L, Becquey E, Kolsteren P, Lachat C, Huybregts L. Fortified Balanced Energy-Protein Supplements Increase Nutrient Adequacy without Displacing Food Intake in Pregnant Women in Rural Burkina Faso. J Nutr. 2021 Dec 3;151(12):3831-3840. doi: 10.1093/jn/nxab289. PMID 34494113
- [Derived] Vanslambrouck K, de Kok B, Toe LC, De Cock N, Ouedraogo M, Dailey-Chwalibog T, Hanley-Cook G, Ganaba R, Lachat C, Huybregts L, Kolsteren P. Effect of balanced energy-protein supplementation during pregnancy and lactation on birth outcomes and infant growth in rural Burkina Faso: study protocol for a randomised controlled trial. BMJ Open. 2021 Mar 24;11(3):e038393. doi: 10.1136/bmjopen-2020-038393. PMID 33762226